CLINICAL TRIAL: NCT02972034
Title: A Phase Ib Study to Evaluate the Safety and Tolerability of MK-8353 in Combination With Pembrolizumab in Patients With Advanced Malignancies
Brief Title: Study of MK-8353 in Combination With Pembrolizumab (MK-3475) in Participants With Advanced Malignancies (MK-8353-013)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: business reasons.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 8353-013; MK-8353-013 (Other: Merck Protocol Number); 2016-003478-42 (EudraCT Number)
Record Dates: First submitted 2016-11-21; First posted 2016-11-23 (Estimated); Results first posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Neoplasms; Colorectal Cancer
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms | interventions — MK-8353; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- A: MK-8353 BID Continuous+Pembro (Experimental): Participants receive MK-8353 orally (PO) two times each day (BID) on Days 1 through 21 of each 21-day cycle PLUS pembrolizumab (pembro) 200 mg intravenously (IV) on Day 1 of each 21-day cycle for up to 35 cycles.
  Interventions: Drug: MK-8353; Biological: Pembrolizumab
- B: MK-8353 QD Continuous+Pembro (Experimental): Participants receive MK-8353 PO once each day (QD) on Days 1 through 21 of each 21-day cycle PLUS pembrolizumab 200 mg IV on Day 1 of each 21-day cycle for up to 35 cycles.
  Interventions: Drug: MK-8353; Biological: Pembrolizumab
- C: MK-8353 QD 1 Week On/1 Week Off+Pembro (Experimental): Optional Arm: Participants receive MK-8353 PO QD on Days 1 to 7, Days 15 to 21 and Days 29 to 35 PLUS pembrolizumab 200 mg IV on Day 1 and Day 22 of each 42-day period (based on 2 cycles of 21 days) for up to 35 cycles.
  Interventions: Drug: MK-8353; Biological: Pembrolizumab
- D: MK-8353 QD Run-in→MK-8353 QD Continuous+Pembro (Experimental): Optional Arm: Participants undergo an MK-8353 PO QD run-in period from Day -14 to Day -1 prior to Cycle 1 during which they receive MK-8353 PO QD. After the run-in period, participants receive MK-8353 PO QD on Days 1 through 21 of each 21-day cycle PLUS pembrolizumab 200 mg IV on Day 1 of each 21-day cycle for up to 36 cycles.
  Interventions: Drug: MK-8353; Biological: Pembrolizumab

INTERVENTIONS:
Drug: MK-8353 — PO capsule
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475

SUMMARY:
This study will evaluate the safety, tolerability and preliminary efficacy of MK-8353 when administered in combination with pembrolizumab (MK-3475). There are two parts in this study: Part 1 will be dose escalation and confirmation, and Part 2 will be a cohort expansion. In Part 1, the recommended phase II dose (RP2D) of MK-8353 in combination with a fixed dose of pembrolizumab in participants with advanced malignancies will be identified and confirmed. Participants will be initially enrolled to receive MK-8353 at 350 mg twice a day (BID) in combination with pembrolizumab at a fixed dose of 200 mg on Day 1 of each 3-week cycle (Q3W) for up to 24 months of treatment. In Part 2, participants with advanced colorectal cancer (CRC) that is microsatellite stable (i.e., non-microsatellite instability-high/deficient mismatch repair [non-MSI-H/dMMR]) who received at least one and up to five prior lines of therapy will be enrolled at the RP2D in the expansion cohort to further evaluate safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Part 1: Has a histologically- or cytologically-documented, locally-advanced or metastatic solid malignancy and has received ≥1 and <6 prior line of cancer treatment regimen(s).
* Part 2: Has a histologically-confirmed adenocarcinoma originating from the colon or rectum (Stage 4 American Joint Committee on Cancer [AJCC] 7th edition) that is microsatellite stable (i.e., non-MSI-H/dMMR). Appendiceal cancer is included AND Has experienced disease progression or was intolerant to at least 1 and up to 5 systemic chemotherapy regimen(s) for metastatic CRC that must have included fluroropyrimidines and irinotecan or oxaliplatin, ± anti-vascular endothelial growth factor (VEGF) or anti-epidermal growth factor receptor (EGFR)(if indicated by RAS mutational status).
* Provides an archival or newly obtained tumor tissue sample and blood samples for biomarker analysis.
* Has ≥1 measurable lesion as defined by RECIST 1.1 on imaging studies.
* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Has adequate organ function
* Female participants of childbearing potential who are willing to use either 2 adequate barrier methods, or to abstain from heterosexual activity throughout the study.
* Male participants of childbearing potential must agree to use an adequate method of contraception.

Exclusion Criteria:

* Has disease that is suitable for local treatment administered with curative intent.
* Part 1: Has received prior therapy with cancer vaccines, or compounds targeting PD-1 (including Merck pembrolizumab [MK-3475]), programmed cell death ligand 1 (PD-L1), PD-L2, cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), or Mitogen-activated protein kinase (MAPK)/Extracellular signal-regulated Kinase (MEK).
* Part 2: Has received prior therapy with cancer vaccines, or compounds targeting PD-1 (including Merck pembrolizumab [MK-3475]), PD-L1, PD-L2, CTLA-4, lymphocyte-activation gene 3 (LAG-3), CD-137, OX-40 (tumor necrosis factor receptor superfamily, member 4 [TNFRSF4], also known as CD134), cluster of differentiation 40 (CD-40), glucocorticoid-induced TNFR-related protein (GITR), serine/threonine-protein kinase B-Raf (BRAF), MEK or other molecules in the MAPK pathway.
* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks prior to the first dose of study drug.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in doses exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has had a prior anticancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or has not recovered (i.e. ≤ Grade 1 or at Baseline) from adverse events (AEs) due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 14 days prior to study Day 1 or who has not recovered (i.e., ≤Grade 1 or at baseline) from AEs due to a previously administered agent.
* Has received transfusion of blood products (including platelets or red blood cells) or administration of colony stimulating factors within 4 weeks prior to study Day 1.
* Has a known additional malignancy that is progressing or requires active treatment.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Has a history of interstitial lung disease.
* Has an active infection requiring systemic therapy.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study.
* Has a known history of Human Immunodeficiency Virus (HIV).
* Has known active Hepatitis B or Hepatitis C.
* Has received a live-virus vaccination within 30 days of planned treatment start.
* Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (3):
- United States (2):
  - Call for Information (Investigational Site 0002), Grand Rapids, Michigan
  - Call for Information (Investigational Site 0001), Nashville, Tennessee
- Merck Canada, Kirkland, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Lakhani NJ, Burris H 3rd, Miller WH Jr, Huang M, Chen LC, Siu LL. A phase 1b study of the ERK inhibitor MK-8353 plus pembrolizumab in patients with advanced solid tumors. Invest New Drugs. 2024 Oct;42(5):581-589. doi: 10.1007/s10637-024-01461-z. Epub 2024 Sep 14. PMID 39276176
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was planned to have two parts. Part 1 was dose escalation and confirmation, and Part 2 was a cohort expansion. The cohort expansion phase (Part 2) was not initiated due to Sponsor's business decision.
Groups:
- Arm A: MK-8353 50 mg + Pembrolizumab: Participants received MK-8353 50 mg orally (PO) two times each day (BID) on Days 1 through 21 of each 21-day cycle PLUS pembrolizumab (pembro) 200 mg intravenously (IV) on Day 1 of each 21-day cycle for up to 35 cycles.
- Arm A: MK-8353 100 mg + Pembrolizumab: Participants received MK-8353 100 mg orally (PO) two times each day (BID) on Days 1 through 21 of each 21-day cycle PLUS pembrolizumab (pembro) 200 mg intravenously (IV) on Day 1 of each 21-day cycle for up to 35 cycles.
- Arm A: MK-8353 50 + 100 mg + Pembrolizumab: Participants received MK-8353 50 mg plus 100 mg orally (PO) two times each day (BID) on Days 1 through 21 of each 21-day cycle PLUS pembrolizumab (pembro) 200 mg intravenously (IV) on Day 1 of each 21-day cycle for up to 35 cycles.
- Arm A: MK-8353 350 mg + Pembrolizumab: Participants received MK-8353 350 mg orally (PO) two times each day (BID) on Days 1 through 21 of each 21-day cycle PLUS pembrolizumab (pembro) 200 mg intravenously (IV) on Day 1 of each 21-day cycle for up to 35 cycles.
- Arm B: MK-8353 50 mg + Pembrolizumab: Participants received MK-8353 PO 50 mg once each day (QD) on Days 1 through 21 of each 21-day cycle PLUS pembrolizumab 200 mg IV on Day 1 of each 21-day cycle for up to 35 cycles.
- Arm B: MK-8353 100 mg + Pembrolizumab: Participants received MK-8353 PO 100 mg once each day (QD) on Days 1 through 21 of each 21-day cycle PLUS pembrolizumab 200 mg IV on Day 1 of each 21-day cycle for up to 35 cycles.
- Arm B: MK-8353 150 mg + Pembrolizumab: Participants received MK-8353 PO 150 mg once each day (QD) on Days 1 through 21 of each 21-day cycle PLUS pembrolizumab 200 mg IV on Day 1 of each 21-day cycle for up to 35 cycles.
- Arm B: MK-8353 200 mg + Pembrolizumab: Participants received MK-8353 PO 200 mg once each day (QD) on Days 1 through 21 of each 21-day cycle PLUS pembrolizumab 200 mg IV on Day 1 of each 21-day cycle for up to 35 cycles.
- Arm B: MK-8353 300 mg + Pembrolizumab: Participants received MK-8353 PO 300 mg once each day (QD) on Days 1 through 21 of each 21-day cycle PLUS pembrolizumab 200 mg IV on Day 1 of each 21-day cycle for up to 35 cycles.
- Arm B: MK-8353 400 mg + Pembrolizumab: Participants received MK-8353 PO 400 mg once each day (QD) on Days 1 through 21 of each 21-day cycle PLUS pembrolizumab 200 mg IV on Day 1 of each 21-day cycle for up to 35 cycles.
- Arm B: MK-8353 600 mg + Pembrolizumab: Participants received MK-8353 PO 600 mg once each day (QD) on Days 1 through 21 of each 21-day cycle PLUS pembrolizumab 200 mg IV on Day 1 of each 21-day cycle for up to 35 cycles.
- Arm C: MK-8353 100 mg + Pembrolizumab: Participants received MK-8353 100 mg PO QD on Days 1 to 7, Days 15 to 21 and Days 29 to 35 PLUS pembrolizumab 200 mg IV on Day 1 and Day 22 of each 42-day period (based on 2 cycles of 21 days) for up to 35 cycles.
- Arm C: MK-8353 150 mg + Pembrolizumab: Participants received MK-8353 150 mg PO QD on Days 1 to 7, Days 15 to 21 and Days 29 to 35 PLUS pembrolizumab 200 mg IV on Day 1 and Day 22 of each 42-day period (based on 2 cycles of 21 days) for up to 35 cycles.
- Arm C: MK-8353 200 mg + Pembrolizumab: Participants received MK-8353 200 mg PO QD on Days 1 to 7, Days 15 to 21 and Days 29 to 35 PLUS pembrolizumab 200 mg IV on Day 1 and Day 22 of each 42-day period (based on 2 cycles of 21 days) for up to 35 cycles.
- Arm C: MK-8353 300 mg + Pembrolizumab: Participants received MK-8353 300 mg PO QD on Days 1 to 7, Days 15 to 21 and Days 29 to 35 PLUS pembrolizumab 200 mg IV on Day 1 and Day 22 of each 42-day period (based on 2 cycles of 21 days) for up to 35 cycles.
Period: Overall Study
Arm/Group | Arm A: MK-8353 50 mg + Pembrolizumab | Arm A: MK-8353 100 mg + Pembrolizumab | Arm A: MK-8353 50 + 100 mg + Pembrolizumab | Arm A: MK-8353 350 mg + Pembrolizumab | Arm B: MK-8353 50 mg + Pembrolizumab | Arm B: MK-8353 100 mg + Pembrolizumab | Arm B: MK-8353 150 mg + Pembrolizumab | Arm B: MK-8353 200 mg + Pembrolizumab | Arm B: MK-8353 300 mg + Pembrolizumab | Arm B: MK-8353 400 mg + Pembrolizumab | Arm B: MK-8353 600 mg + Pembrolizumab | Arm C: MK-8353 100 mg + Pembrolizumab | Arm C: MK-8353 150 mg + Pembrolizumab | Arm C: MK-8353 200 mg + Pembrolizumab | Arm C: MK-8353 300 mg + Pembrolizumab
Started | 14 | 1 | 3 | 4 | 4 | 3 | 4 | 7 | 10 | 14 | 8 | 3 | 14 | 11 | 11
Treated | 14 | 1 | 3 | 4 | 4 | 3 | 4 | 7 | 10 | 14 | 8 | 3 | 13 | 11 | 11
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 14 | 1 | 3 | 4 | 4 | 3 | 4 | 7 | 10 | 14 | 8 | 3 | 14 | 11 | 11
Not completed — Death | 11 | 1 | 3 | 3 | 2 | 2 | 3 | 4 | 8 | 11 | 3 | 2 | 11 | 10 | 9
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 2 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 1 | 0
Not completed — Screen Failure | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population consisted of all participants who received received at least 1 dose of study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: MK-8353 50 mg + Pembrolizumab | Arm A: MK-8353 100 mg + Pembrolizumab | Arm A: MK-8353 50 + 100 mg + Pembrolizumab | Arm A: MK-8353 350 mg + Pembrolizumab | Arm B: MK-8353 50 mg + Pembrolizumab | Arm B: MK-8353 100 mg + Pembrolizumab | Arm B: MK-8353 150 mg + Pembrolizumab | Arm B: MK-8353 200 mg + Pembrolizumab | Arm B: MK-8353 300 mg + Pembrolizumab | Arm B: MK-8353 400 mg + Pembrolizumab | Arm B: MK-8353 600 mg + Pembrolizumab | Arm C: MK-8353 100 mg + Pembrolizumab | Arm C: MK-8353 150 mg + Pembrolizumab | Arm C: MK-8353 200 mg + Pembrolizumab | Arm C: MK-8353 300 mg + Pembrolizumab | Total
Number analyzed (Participants) | 14 | 1 | 3 | 4 | 4 | 3 | 4 | 7 | 10 | 14 | 8 | 3 | 14 | 11 | 11 | 111
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.8 (10.1) | 51.0 (NA) — Method of dispersion could not be estimated due to N=1 | 59.7 (13.0) | 46.0 (8.7) | 57.5 (11.1) | 60.0 (14.5) | 57.5 (6.2) | 63.1 (8.5) | 61.1 (10.3) | 59.5 (8.1) | 62.1 (11.6) | 58.0 (19.3) | 53.0 (8.9) | 64.1 (8.2) | 57.6 (12.8) | 58.3 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 2 | 1 | 2 | 0 | 2 | 4 | 2 | 5 | 5 | 3 | 8 | 2 | 7 | 49
  Male | 9 | 0 | 1 | 3 | 2 | 3 | 2 | 3 | 8 | 9 | 3 | 0 | 6 | 9 | 4 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 1 | 2 | 4 | 3 | 3 | 2 | 4 | 8 | 12 | 8 | 3 | 12 | 11 | 9 | 94
  Unknown or Not Reported | 2 | 0 | 1 | 0 | 1 | 0 | 2 | 3 | 2 | 2 | 0 | 0 | 2 | 0 | 2 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 3 | 2 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 3
  White | 14 | 1 | 3 | 4 | 4 | 3 | 3 | 5 | 9 | 13 | 6 | 3 | 12 | 8 | 7 | 95
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 4
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Participants in the study were required to have an ECOG Performance Status of 0 (Fully active, able to carry on all pre-disease performance without restriction) or 1 (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature). The analysis population consisted of all participants who received received at least 1 dose of study intervention.
  Participants
    ECOG = 0 | 5 | 0 | 0 | 2 | 2 | 1 | 0 | 4 | 2 | 7 | 1 | 2 | 6 | 3 | 6 | 41
    ECOG = 1 | 9 | 1 | 3 | 2 | 2 | 2 | 4 | 3 | 8 | 7 | 7 | 1 | 7 | 8 | 5 | 69
    Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: Number of participants who experienced an AE was defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study therapy and irrespective of causality to study treatment
Time Frame: Up to 27 months
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: MK-8353 50 mg + Pembrolizumab | Arm A: MK-8353 100 mg + Pembrolizumab | Arm A: MK-8353 50 + 100 mg + Pembrolizumab | Arm A: MK-8353 350 mg + Pembrolizumab | Arm B: MK-8353 50 mg + Pembrolizumab | Arm B: MK-8353 100 mg + Pembrolizumab | Arm B: MK-8353 150 mg + Pembrolizumab | Arm B: MK-8353 200 mg + Pembrolizumab | Arm B: MK-8353 300 mg + Pembrolizumab | Arm B: MK-8353 400 mg + Pembrolizumab | Arm B: MK-8353 600 mg + Pembrolizumab | Arm C: MK-8353 100 mg + Pembrolizumab | Arm C: MK-8353 150 mg + Pembrolizumab | Arm C: MK-8353 200 mg + Pembrolizumab | Arm C: MK-8353 300 mg + Pembrolizumab
Number analyzed (Participants) | 14 | 1 | 3 | 4 | 4 | 3 | 4 | 7 | 10 | 14 | 8 | 3 | 13 | 11 | 11
Participants | 14 | 1 | 3 | 4 | 4 | 3 | 4 | 7 | 10 | 14 | 8 | 3 | 13 | 11 | 11

2. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinued treatment due to an AE was assessed.
Time Frame: Up to 24 months
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: MK-8353 50 mg + Pembrolizumab | Arm A: MK-8353 100 mg + Pembrolizumab | Arm A: MK-8353 50 + 100 mg + Pembrolizumab | Arm A: MK-8353 350 mg + Pembrolizumab | Arm B: MK-8353 50 mg + Pembrolizumab | Arm B: MK-8353 100 mg + Pembrolizumab | Arm B: MK-8353 150 mg + Pembrolizumab | Arm B: MK-8353 200 mg + Pembrolizumab | Arm B: MK-8353 300 mg + Pembrolizumab | Arm B: MK-8353 400 mg + Pembrolizumab | Arm B: MK-8353 600 mg + Pembrolizumab | Arm C: MK-8353 100 mg + Pembrolizumab | Arm C: MK-8353 150 mg + Pembrolizumab | Arm C: MK-8353 200 mg + Pembrolizumab | Arm C: MK-8353 300 mg + Pembrolizumab
Number analyzed (Participants) | 14 | 1 | 3 | 4 | 4 | 3 | 4 | 7 | 10 | 14 | 8 | 3 | 13 | 11 | 11
Participants | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 4 | 2 | 0 | 3 | 2 | 0

3. Primary Outcome: Number of Participants Who Experienced Dose-Limiting Toxicity (DLT)
Description: DLT was defined as a treatment-related adverse event (AE) including the following: Grade (Gr) 4 nonhematologic toxicity (not laboratory), Gr 4 hematologic toxicity lasting ≥7 days, except thrombocytopenia or Gr 4 thrombocytopenia of any duration or Gr 3 thrombocytopenia associated with clinically significant bleeding, Gr 3 non-hematological AE with the exception of fatigue lasting >3 days despite optimal supportive care, any Gr 3 or Gr 4 nonhematologic laboratory value if medical intervention is required to treat the subject, or abnormality leads to hospitalization or abnormality persists for >1 week, Gr 3 or Gr 4 febrile neutropenia, prolonged delay (>2 weeks) in initiating Cycle 2 due to treatment-related toxicity, any treatment-related toxicity that causes the subject to discontinue treatment during Cycle 1, missing >25% of MK-8353 doses as a result of drug-related AE(s) during the first cycle, Gr 5 toxicity.
Time Frame: Cycle 1 (Arms A, B & C: Up to 21 days)
Population: The DLT evaluable population consisted of all participants who completed the first cycle of study treatment or who discontinued from the study due to a drug-related AE.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: MK-8353 50 mg + Pembrolizumab | Arm A: MK-8353 100 mg + Pembrolizumab | Arm A: MK-8353 50 + 100 mg + Pembrolizumab | Arm A: MK-8353 350 mg + Pembrolizumab | Arm B: MK-8353 50 mg + Pembrolizumab | Arm B: MK-8353 100 mg + Pembrolizumab | Arm B: MK-8353 150 mg + Pembrolizumab | Arm B: MK-8353 200 mg + Pembrolizumab | Arm B: MK-8353 300 mg + Pembrolizumab | Arm B: MK-8353 400 mg + Pembrolizumab | Arm B: MK-8353 600 mg + Pembrolizumab | Arm C: MK-8353 100 mg + Pembrolizumab | Arm C: MK-8353 150 mg + Pembrolizumab | Arm C: MK-8353 200 mg + Pembrolizumab | Arm C: MK-8353 300 mg + Pembrolizumab
Number analyzed (Participants) | 13 | 1 | 3 | 4 | 4 | 3 | 4 | 7 | 7 | 13 | 7 | 3 | 12 | 9 | 10
Participants | 0 | 1 | 2 | 3 | 0 | 0 | 0 | 1 | 0 | 4 | 3 | 0 | 2 | 1 | 2

4. Secondary Outcome: Objective Response Rate (ORR) Based on Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by the Investigator
Description: ORR was defined as the percentage of the participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters). The ORR per RECIST 1.1 as assessed by Investigator was presented.
Time Frame: Up to 24 months
Population: Analysis population consisted of all participants who had a baseline scan with measurable disease by investigator assessment and who were administered a dose of the study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm A: MK-8353 50 mg + Pembrolizumab | Arm A: MK-8353 100 mg + Pembrolizumab | Arm A: MK-8353 50 + 100 mg + Pembrolizumab | Arm A: MK-8353 350 mg + Pembrolizumab | Arm B: MK-8353 50 mg + Pembrolizumab | Arm B: MK-8353 100 mg + Pembrolizumab | Arm B: MK-8353 150 mg + Pembrolizumab | Arm B: MK-8353 200 mg + Pembrolizumab | Arm B: MK-8353 300 mg + Pembrolizumab | Arm B: MK-8353 400 mg + Pembrolizumab | Arm B: MK-8353 600 mg + Pembrolizumab | Arm C: MK-8353 100 mg + Pembrolizumab | Arm C: MK-8353 150 mg + Pembrolizumab | Arm C: MK-8353 200 mg + Pembrolizumab | Arm C: MK-8353 300 mg + Pembrolizumab
Number analyzed (Participants) | 14 | 1 | 3 | 4 | 4 | 3 | 4 | 7 | 10 | 14 | 8 | 3 | 13 | 11 | 11
Percentage of Participants | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 97.5] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 41.0] | 20.0 [2.5 to 55.6] | 21.4 [4.7 to 50.8] | 25.0 [3.2 to 65.1] | 0.0 [0.0 to 70.8] | 7.7 [0.2 to 36.0] | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 28.5]

5. Secondary Outcome: Percent Change in Cancer Antigen 125 (CA-125)
Description: CA-125 was the tumour biomarker used to test cancer. Disease progression is indicated by CA-125 tumor marker elevation.
Time Frame: Cycle 1-8 Day 1, and end of treatment/ safety follow-up (30 days after the last dose). Each cycle was 21 days.
Population: Analysis population consisted of all participants who had a baseline scan with measurable disease by investigator assessment, CA-125 data available for each timepoint and who were administered a dose of the study treatment.
Measure: Mean (Full Range); unit: Percent Change
Arm/Group | Arm A: MK-8353 50 mg + Pembrolizumab | Arm A: MK-8353 100 mg + Pembrolizumab | Arm A: MK-8353 50 + 100 mg + Pembrolizumab | Arm A: MK-8353 350 mg + Pembrolizumab | Arm B: MK-8353 50 mg + Pembrolizumab | Arm B: MK-8353 100 mg + Pembrolizumab | Arm B: MK-8353 150 mg + Pembrolizumab | Arm B: MK-8353 200 mg + Pembrolizumab | Arm B: MK-8353 300 mg + Pembrolizumab | Arm B: MK-8353 400 mg + Pembrolizumab | Arm B: MK-8353 600 mg + Pembrolizumab | Arm C: MK-8353 100 mg + Pembrolizumab | Arm C: MK-8353 150 mg + Pembrolizumab | Arm C: MK-8353 200 mg + Pembrolizumab | Arm C: MK-8353 300 mg + Pembrolizumab
Number analyzed (Participants) | 3 | 0 | 1 | 0 | 1 | 1 | 2 | 4 | 1 | 2 | 2 | 1 | 1 | 0 | 5
Percent Change
  Day 1 Cycle 2: number analyzed (Participants) | 3 | 0 | 1 | 0 | 1 | 1 | 2 | 4 | 0 | 0 | 2 | 1 | 1 | 0 | 5
  Day 1 Cycle 2 | 15.47 [-15.2 to 56.7] |  | 17.2 [17.2 to 17.2] |  | -13.3 [-13.3 to -13.3] | 68.3 [68.3 to 68.3] | 83.75 [-9.3 to 176.8] | 39.85 [0.0 to 137.2] |  |  | 11.00 [-75.8 to 97.8] | 367.6 [367.6 to 367.6] | -60.00 [-60.0 to -60.0] |  | 36.36 [-11.8 to 112.5]
  Day 1 Cycle 3: number analyzed (Participants) | 3 | 0 | 1 | 0 | 1 | 0 | 2 | 4 | 0 | 0 | 2 | 1 | 1 | 0 | 2
  Day 1 Cycle 3 | 42.69 [-27.3 to 80.0] |  | 33.0 [33.0 to 33.0] |  | -13.3 [-13.3 to -13.3] |  | -31.21 [-46.4 to -16.0] | 80.55 [11.1 to 221.8] |  |  | 262.56 [-87.9 to 613.0] | 300.3 [300.3 to 300.3] | -78.8 [-78.8 to -78.8] |  | -5.10 [-23.5 to 13.3]
  Day 1 Cycle 4: number analyzed (Participants) | 2 | 0 | 0 | 0 | 1 | 0 | 2 | 3 | 0 | 0 | 0 | 1 | 1 | 0 | 2
  Day 1 Cycle 4 | 103.10 [96.7 to 109.5] |  |  |  | -13.3 [-13.3 to -13.3] |  | -24.19 [-71.4 to 23.0] | 42.26 [0.0 to 87.5] |  |  |  | 359.1 [359.1 to 359.1] | -78.8 [-78.8 to -78.8] |  | -10.05 [-11.8 to -8.3]
  Day 1 Cycle 5: number analyzed (Participants) | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0
  Day 1 Cycle 5 | 153.25 [70.0 to 236.5] |  |  |  | -13.3 [-13.3 to -13.3] |  | -76.8 [-76.8 to -76.8] | 22.2 [22.2 to 22.2] |  |  | -88.89 [-88.89 to -88.89] | 451.9 [451.9 to 451.9] | -82.4 [-82.4 to -82.4] |  |
  Day 1 Cycle 6: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
  Day 1 Cycle 6 | 50.0 [50.0 to 50.0] |  |  |  | -6.7 [-6.7 to -6.7] |  | -75.0 [-75.0 to -75.0] |  |  |  | -88.89 [-88.89 to -88.89] |  | -87.1 [-87.1 to -87.1] |  | -25.0 [-25.0 to -25.0]
  Day 1 Cycle 7: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
  Day 1 Cycle 7 | 36.7 [36.7 to 36.7] |  |  |  |  |  |  |  |  |  | -89.9 [-89.9 to -89.9] |  | -84.7 |  | -16.7
  Day 1 Cycle 8: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Day 1 Cycle 8 | 3.3 [3.3 to 3.3] |  |  |  |  |  |  |  |  |  | -90.9 [-90.9 to -90.9] |  |  |  | -16.7 [-16.7 to -16.7]
  End of treatment/ Safety Follow-up: number analyzed (Participants) | 2 | 0 | 1 | 0 | 0 | 1 | 2 | 2 | 1 | 2 | 2 | 0 | 0 | 0 | 5
  End of treatment/ Safety Follow-up | 118.18 [-36.7 to 273.0] |  | 101.7 [101.7 to 101.7] |  |  | 329.3 [329.3 to 329.3] | 2.69 [-76.8 to 82.2] | 256.48 [157.1 to 355.8] | 38.6 [38.6 to 38.6] | 695.94 [164.3 to 1227.6] | -30.24 [-89.9 to 29.4] |  |  |  | 87.88 [-11.8 to 376.9]

6. Secondary Outcome: Percent Change in Carcinoembryonic Antigen (CEA)
Description: CEA was the tumour biomarker used to test cancer. Disease progression is indicated by CEA tumor marker elevation.
Time Frame: Cycle 1-9 Day 1, and end of treatment/ safety follow-up (30 days after the last dose). Each cycle was 21 days
Population: Analysis population consisted of all participants who had a baseline scan with measurable disease by investigator assessment, CEA data available for each timepoint and who were administered a dose of the study treatment.
Measure: Mean (Full Range); unit: Percent Change
Arm/Group | Arm A: MK-8353 50 mg + Pembrolizumab | Arm A: MK-8353 100 mg + Pembrolizumab | Arm A: MK-8353 50 + 100 mg + Pembrolizumab | Arm A: MK-8353 350 mg + Pembrolizumab | Arm B: MK-8353 50 mg + Pembrolizumab | Arm B: MK-8353 100 mg + Pembrolizumab | Arm B: MK-8353 150 mg + Pembrolizumab | Arm B: MK-8353 200 mg + Pembrolizumab | Arm B: MK-8353 300 mg + Pembrolizumab | Arm B: MK-8353 400 mg + Pembrolizumab | Arm B: MK-8353 600 mg + Pembrolizumab | Arm C: MK-8353 100 mg + Pembrolizumab | Arm C: MK-8353 150 mg + Pembrolizumab | Arm C: MK-8353 200 mg + Pembrolizumab | Arm C: MK-8353 300 mg + Pembrolizumab
Number analyzed (Participants) | 10 | 1 | 1 | 2 | 3 | 2 | 1 | 3 | 2 | 4 | 2 | 3 | 5 | 3 | 5
Percent Change
  Day 1 Cycle 2: number analyzed (Participants) | 10 | 0 | 1 | 2 | 3 | 2 | 1 | 3 | 2 | 4 | 2 | 3 | 5 | 3 | 5
  Day 1 Cycle 2 | 2.08 [-64.4 to 83.0] |  | 8.3 [8.3 to 8.3] | -0.27 [-17.2 to 16.7] | 54.41 [26.9 to 81.5] | -6.72 [-16.7 to 3.2] | -80.1 [-80.1 to -80.1] | -13.8 [-38.4 to 4.9] | 21.6 [21.6 to 21.6] | 46.01 [4.9 to 66.8] | 18.68 [16.7 to 20.7] | 7.75 [-6.3 to 22.4] | 47.43 [-12.2 to 204.2] | 58.20 [34.6 to 91.2] | 62.24 [-18.8 to 172.5]
  Day 1 Cycle 3: number analyzed (Participants) | 9 | 0 | 1 | 0 | 3 | 0 | 1 | 3 | 2 | 0 | 2 | 2 | 5 | 1 | 4
  Day 1 Cycle 3 | 45.35 [-37.1 to 162.8] |  | 5.6 [5.6 to 5.6] |  | 113.63 [66.2 to 161.3] |  | -93.9 [-93.9 to -93.9] | 4.86 [-18.5 to 33.1] | 9.0 [9.0 to 9.0] |  | 66.7 [66.7 to 66.7] | 35.17 [31.3 to 39.1] | 129.52 [-10.5 to 525.0] | 23.8 [23.8 to 23.8] | 129.98 [-18.8 to 316.0]
  Day 1 Cycle 4: number analyzed (Participants) | 4 | 0 | 0 | 1 | 2 | 0 | 1 | 2 | 2 | 4 | 0 | 2 | 4 | 1 | 1
  Day 1 Cycle 4 | -1.84 [-26.7 to 42.9] |  |  | 50.0 [50.0 to 50.0] | 199.86 [90.0 to 309.7] |  | -95.1 [-95.1 to -95.1] | 19.07 [6.7 to 31.5] | -38.1 [-38.1 to -38.1] | 17.6 [17.6 to 17.6] |  | 178.49 [25.0 to 332.0] | 36.58 [-10.5 to 91.7] | -51.1 [-51.1 to -51.1] | 315.8 [315.8 to 315.8]
  Day 1 Cycle 5: number analyzed (Participants) | 3 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 3 | 1 | 0
  Day 1 Cycle 5 | -8.08 [-39.5 to 28.6] |  |  | 66.67 [66.67 to 66.67] | 197.72 [63.2 to 332.3] |  | -96.5 [-96.5 to -96.5] | 106.6 [106.6 to 106.6] | -44.2 [-44.2 to -44.2] |  |  | 50.00 [50.00 to 50.00] | 42.31 [-15.8 to 82.7] | -67.8 [-67.8 to -67.8] |
  Day 1 Cycle 6: number analyzed (Participants) | 2 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0
  Day 1 Cycle 6 | 2.88 [-2.88 to 28.6] |  |  | 61.1 [61.1 to 61.1] | 445.2 [445.2 to 445.2] |  | -96.6 [-96.6 to -96.6] |  |  | 29.4 [29.4 to 29.4] |  |  | 24.7 [-21.1 to 70.0] | -35.8 [-35.8 to -35.8] |
  Day 1 Cycle 7: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Day 1 Cycle 7 | 29.64 [28.6 to 30.7] |  |  |  |  |  |  |  |  |  |  |  | 70.0 [70.0 to 70.0] |  |
  Day 1 Cycle 8: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Day 1 Cycle 8 | 27.01 [25.4 to 28.6] |  |  |  |  |  |  |  |  | 0.00 [0.00 to 0.00] |  |  |  |  |
  Day 1 Cycle 9: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Day 1 Cycle 9 | 28.6 [28.6 to 28.6] |  |  |  |  |  |  |  |  | 23.5 [23.5 to 23.5] |  |  |  |  |
  End of treatment/ Safety Follow-up: number analyzed (Participants) | 6 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 2 | 3 | 2 | 0 | 3 | 2 | 5
  End of treatment/ Safety Follow-up | 46.99 [-12.3 to 153.8] | 200.00 [200.00 to 200.00] | -2.8 [-2.8 to -2.8] | -79.1 [-79.1 to -79.1] | 232.8 [232.8 to 232.8] | 108.3 [108.3 to 108.3] | -93.7 [-93.7 to -93.7] |  | 84.85 [52.7 to 117.0] | -7.67 [-17.6 to 9.1] | 56.51 [-11.1 to 124.1] |  | 58.14 [-7.3 to 141.7] | 42.64 [-13.9 to 99.2] | 416.18 [-6.3 to 1430.2]

7. Secondary Outcome: Percent Change in Carbohydrate Antigen (CA19-9)
Description: CA19-9 was the tumour biomarker used to test cancer. Disease progression is indicated by CA19-9 tumor marker elevation
Time Frame: Cycle 1-7 Day 1, and end of treatment/ safety follow-up (30 days after the last dose). Each cycle was 21 days.
Population: Analysis population consisted of all participants who had a baseline scan with measurable disease by investigator assessment, CA19-9 data available for each timepoint and who were administered a dose of the study treatment.
Measure: Mean (Full Range); unit: Percent Change
Arm/Group | Arm A: MK-8353 50 mg + Pembrolizumab | Arm A: MK-8353 100 mg + Pembrolizumab | Arm A: MK-8353 50 + 100 mg + Pembrolizumab | Arm A: MK-8353 350 mg + Pembrolizumab | Arm B: MK-8353 50 mg + Pembrolizumab | Arm B: MK-8353 100 mg + Pembrolizumab | Arm B: MK-8353 150 mg + Pembrolizumab | Arm B: MK-8353 200 mg + Pembrolizumab | Arm B: MK-8353 300 mg + Pembrolizumab | Arm B: MK-8353 400 mg + Pembrolizumab | Arm B: MK-8353 600 mg + Pembrolizumab | Arm C: MK-8353 100 mg + Pembrolizumab | Arm C: MK-8353 150 mg + Pembrolizumab | Arm C: MK-8353 200 mg + Pembrolizumab | Arm C: MK-8353 300 mg + Pembrolizumab
Number analyzed (Participants) | 4 | 0 | 2 | 0 | 1 | 2 | 1 | 3 | 3 | 2 | 4 | 1 | 3 | 3 | 4
Percent Change
  Day 1 Cycle 2 | 36.10 [-21.4 to 95.8] |  | -2.06 [-7.7 to 3.6] |  | 12.2 [12.2 to 12.2] | 51.34 [23.2 to 79.5] | -73.9 [-73.9 to -73.9] | 19.93 [-8.3 to 57.0] | 64.28 [-61.6 to 190.2] | 0.9 [0.9 to 0.9] | -8.23 [-97.1 to 80.6] | 12.5 [12.5 to 12.5] | 100.88 [-14.6 to 242.3] | -5.3 [-5.3 to -5.3] | 240.00 [-15.4 to 811.9]
  Day 1 Cycle 3: number analyzed (Participants) | 3 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 3 | 0 | 4 | 1 | 3 | 3 | 3
  Day 1 Cycle 3 | 44.52 [3.6 to 80.0] |  | -23.1 [-23.1 to -23.1] |  | 71.6 [71.6 to 71.6] | 63.4 [63.4 to 63.4] | 78.3 [78.3 to 78.3] | 1.39 [-22.2 to 25.0] | 189.69 [-93.8 to 473.2] |  | 514.26 [-98.0 to 1126.6] | 25.0 [25.0 to 25.0] | 119.07 [-30.6 to 362.8] | -15.8 [-15.8 to -15.8] | 799.42 [-15.4 to 2153.9]
  Day 1 Cycle 4: number analyzed (Participants) | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 0 | 1 | 1 | 2 | 3 | 1
  Day 1 Cycle 4 | 40.48 [16.7 to 64.3] |  |  |  | 168.9 [168.9 to 168.9] | 199.1 [199.1 to 199.1] | -73.9 [-73.9 to -73.9] | 43.06 [11.1 to 75.0] | -91.1 [-91.1 to -91.1] |  | -98.8 [-98.8 to -98.8] | 75.0 [75.0 to 75.0] | 29.24 [25.0 to 33.5] | 10.5 [10.5 to 10.5] | 450.7 [450.7 to 450.7]
  Day 1 Cycle 5: number analyzed (Participants) | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 3 | 0
  Day 1 Cycle 5 | 113.10 [33.3 to 192.9] |  |  |  | 168.9 [168.9 to 168.9] | 81.3 [81.3 to 81.3] | -78.3 [-78.3 to -78.3] | 206.3 [206.3 to 206.3] | 1346.4 [1346.4 to 1346.4] |  | -99.0 [-99.0 to -99.0] | 150.0 [150.0 to 150.0] | 50.0 [50.0 to 50.0] | -5.3 [-5.3 to -5.3] |
  Day 1 Cycle 6: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Day 1 Cycle 6 | 16.7 [16.7 to 16.7] |  |  |  | 202.7 [202.7 to 202.7] |  | -73.9 [-73.9 to -73.9] |  |  |  |  | 25.00 [25.00 to 25.00] | -10.5 [-10.5 to -10.5] |  |
  Day 1 Cycle 7: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Day 1 Cycle 7 | 33.33 [33.33 to 33.33] |  |  |  |  |  |  |  |  |  | -99.1 [-99.1 to -99.1] |  | 50.0 [50.0 to 50.0] |  |
  End of treatment/ Safety Follow-up: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 2 | 4 | 0 | 2 | 3 | 3
  End of treatment/ Safety Follow-up | 89.29 [0.0 to 178.6] |  |  |  |  | -99.5 [-99.5 to -99.5] | -71.7 [-71.7 to -71.7] |  | 1078.56 [-91.4 to 3177.1] | -4.70 [-47.9 to 38.5] | 850.28 [-99.5 to 3413.1] |  | 538.54 [277.1 to 800.0] | 54.42 [-2.5 to 139.5] | 11152.37 [55.6 to 32853.8]

ADVERSE EVENTS:
Time Frame: Up to ~ 27 months
Description: All-cause mortality includes all allocated participants. AEs include participants who received ≥1 dose of study treatment. Per protocol, disease progression was not considered an AE, unless related to study treatment. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study treatment were excluded as AEs.
Arm/Group | Arm A: MK-8353 50 mg + Pembrolizumab | Arm A: MK-8353 100 mg + Pembrolizumab | Arm A: MK-8353 50 + 100 mg + Pembrolizumab | Arm A: MK-8353 350 mg + Pembrolizumab | Arm B: MK-8353 50 mg + Pembrolizumab | Arm B: MK-8353 100 mg + Pembrolizumab | Arm B: MK-8353 150 mg + Pembrolizumab | Arm B: MK-8353 200 mg + Pembrolizumab | Arm B: MK-8353 300 mg + Pembrolizumab | Arm B: MK-8353 400 mg + Pembrolizumab | Arm B: MK-8353 600 mg + Pembrolizumab | Arm C: MK-8353 100 mg + Pembrolizumab | Arm C: MK-8353 150 mg + Pembrolizumab | Arm C: MK-8353 200 mg + Pembrolizumab | Arm C: MK-8353 300 mg + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 13/14 | 1/1 | 3/3 | 3/4 | 3/4 | 2/3 | 3/4 | 4/7 | 8/10 | 11/14 | 5/8 | 3/3 | 11/14 | 10/11 | 9/11
Serious Adverse Events (participants affected / at risk) | 6/14 | 1/1 | 0/3 | 3/4 | 1/4 | 1/3 | 2/4 | 1/7 | 3/10 | 3/14 | 5/8 | 1/3 | 5/13 | 4/11 | 4/11
Other Adverse Events (participants affected / at risk) | 14/14 | 1/1 | 3/3 | 4/4 | 4/4 | 3/3 | 4/4 | 7/7 | 10/10 | 14/14 | 8/8 | 3/3 | 13/13 | 11/11 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: MK-8353 50 mg + Pembrolizumab (N=14) | Arm A: MK-8353 100 mg + Pembrolizumab (N=1) | Arm A: MK-8353 50 + 100 mg + Pembrolizumab (N=3) | Arm A: MK-8353 350 mg + Pembrolizumab (N=4) | Arm B: MK-8353 50 mg + Pembrolizumab (N=4) | Arm B: MK-8353 100 mg + Pembrolizumab (N=3) | Arm B: MK-8353 150 mg + Pembrolizumab (N=4) | Arm B: MK-8353 200 mg + Pembrolizumab (N=7) | Arm B: MK-8353 300 mg + Pembrolizumab (N=10) | Arm B: MK-8353 400 mg + Pembrolizumab (N=14) | Arm B: MK-8353 600 mg + Pembrolizumab (N=8) | Arm C: MK-8353 100 mg + Pembrolizumab (N=3) | Arm C: MK-8353 150 mg + Pembrolizumab (N=13) | Arm C: MK-8353 200 mg + Pembrolizumab (N=11) | Arm C: MK-8353 300 mg + Pembrolizumab (N=11)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacillus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Schizophrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: MK-8353 50 mg + Pembrolizumab (N=14) | Arm A: MK-8353 100 mg + Pembrolizumab (N=1) | Arm A: MK-8353 50 + 100 mg + Pembrolizumab (N=3) | Arm A: MK-8353 350 mg + Pembrolizumab (N=4) | Arm B: MK-8353 50 mg + Pembrolizumab (N=4) | Arm B: MK-8353 100 mg + Pembrolizumab (N=3) | Arm B: MK-8353 150 mg + Pembrolizumab (N=4) | Arm B: MK-8353 200 mg + Pembrolizumab (N=7) | Arm B: MK-8353 300 mg + Pembrolizumab (N=10) | Arm B: MK-8353 400 mg + Pembrolizumab (N=14) | Arm B: MK-8353 600 mg + Pembrolizumab (N=8) | Arm C: MK-8353 100 mg + Pembrolizumab (N=3) | Arm C: MK-8353 150 mg + Pembrolizumab (N=13) | Arm C: MK-8353 200 mg + Pembrolizumab (N=11) | Arm C: MK-8353 300 mg + Pembrolizumab (N=11)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Ascites (Gastrointestinal disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 2 (2) | 3 (3) | 4 (9) | 2 (2) | 5 (7) | 2 (2) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 5 (6) | 4 (4) | 1 (1) | 2 (2) | 5 (5) | 3 (5) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5) | 0 (0) | 0 (0) | 2 (3) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 5 (12) | 3 (3) | 1 (2) | 2 (2) | 2 (3) | 3 (4) | 1 (1)
Asthenia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 2 (3) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 5 (5) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 4 (4) | 8 (8) | 3 (3) | 2 (2) | 2 (2) | 4 (4) | 2 (2)
Oedema peripheral (General disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (8) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (2) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (6) | 3 (4) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 3 (4) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 3 (6) | 2 (7) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 2 (3) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 3 (4) | 2 (6) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 2 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 4 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 3 (3) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abnormal faeces (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tongue discolouration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ill-defined disorder (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Portal hypertension (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess neck (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adjusted calcium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood magnesium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema genital (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scrotal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scrotal swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypohidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Umbilical discharge (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/34/NCT02972034/Prot_SAP_000.pdf